CLINICAL TRIAL: NCT01197794
Title: A Double-blind, Placebo-controlled, Randomised, Parallel-group, Phase II, Multi-centre Study to Assess the Efficacy, Safety and Tolerability of 4 Twice Daily Doses and 2 Once Daily Doses of AZD1981 Given as Tablets During 12 Weeks in Asthmatic Patients
Brief Title: Investigation of Efficacy, Safety and Tolerability of Once and Twice Daily Doses of AZD1981 in Asthmatic Patients
Acronym: Sweapea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9830C00008; 2010-020407-73 (EudraCT Number)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2013-09-10 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Asthma Patients
Keywords: Efficacy; safety; tolerability; dose finding; asthma patients
MeSH Terms: interventions — AZD1981

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- AZD1981 10 mg (Experimental): AZD1981 10 mg
  Interventions: Drug: AZD1981
- AZD1981 40 mg (Experimental): AZD1981 40 mg
  Interventions: Drug: AZD1981
- AZD1981 100 mg (Experimental): AZD1981 100 mg
  Interventions: Drug: AZD1981
- AZD1981 400 mg (Experimental): AZD1981 400 mg
  Interventions: Drug: AZD1981
- AZD1981 80 mg (Experimental): AZD1981 80 mg
  Interventions: Drug: AZD1981
- AZD1981 200 mg (Experimental): AZD1981 200 mg
  Interventions: Drug: AZD1981
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1981 — AZD1981 twice daily
  Arms: AZD1981 10 mg; AZD1981 100 mg; AZD1981 40 mg; AZD1981 400 mg
Drug: AZD1981 — AZD1981 once daily
  Arms: AZD1981 200 mg; AZD1981 80 mg
Drug: Placebo — Placebo to match AZD1981
  Arms: Placebo

SUMMARY:
The study will assess the efficacy, safety and tolerability of AZD1981 compared to non-active compound in asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women. Women must be surgically sterilized/postmenopausal or use double barrier method contraception
* 6 months history of asthma according to ATS definition
* Prescribed daily dose of ICS and LABA for at least 3 months prior to Visit 2
* Pre-bronchodilator FEV1 of 40 to 85 % of predicted normal
* A total ACQ5 score of 1.5 or more

Exclusion Criteria:

* Respiratory infection significantly affecting the asthma
* Any significant disease and disorder that may put the patient at risk or influence study results
* Any clinically relevant abnormal findings
* A smoking history of more than 10 pack years
* Intake of oral, rectal or parenteral glucocorticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1144 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, Study Director — AstraZeneca
Locations (105):
- United States (19):
  - Research Site, Fullerton, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Wheaton, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Bellevue, Nebraska
  - Research Site, Sylvania, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Collegeville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Clinton, South Carolina
  - Research Site, Waco, Texas
  - Research Site, Tacoma, Washington
- Argentina (5):
  - Research Site, Buenos Aires, Argentina
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Mendoza, Mendoza Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
- Brazil (8):
  - Research Site, Porto Alegre, Brasil
  - Research Site, Vitória, Espírito Santo
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Juiz de Fora, Minas Gerais
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Florian Polis, Santa Catarina
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
- Japan (26):
  - Research Site, Yanagawa, Fukuoka
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Chitose, Hokkaido
  - Research Site, Kitahiroshima, Hokkaido
  - Research Site, Obihiro, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tomakomai, Hokkaido
  - Research Site, Himeji, Hyōgo
  - Research Site, Naka-gun, Ibaraki
  - Research Site, Sakaidechō, Kagawa-ken
  - Research Site, Fujisawa-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kochi, Kochi
  - Research Site, Kyoto, Kyoto
  - Research Site, Nagaoka, Niigata
  - Research Site, Beppu, Oita Prefecture
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Kurashiki-shi, Okayama-ken
  - Research Site, Matsue, Shimane
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Chūō, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Kodaira, Tokyo
  - Research Site, Nakano-ku, Tokyo
  - Research Site, Ohota-ku, Tokyo
- Mexico (5):
  - Research Site, México, D.f.
  - Research Site, Tijuana, Estado de Baja California
  - Research Site, Morelia, Michoacán
  - Research Site, Monterrey, Nuevo León
  - Research Site, Guadalajara
- Romania (6):
  - Research Site, Constanța, Constanța County
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Iași
  - Research Site, Tg. Mures
- Russia (5):
  - Research Site, Moscow, Russia
  - Research Site, Yekaterinburg, Russia
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Vladikavkaz
- Slovakia (15):
  - Research Site, Banská Bystrica
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Dunajská Streda
  - Research Site, Hnúšťa
  - Research Site, Komárno
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Liptovský Hrádok
  - Research Site, Liptovský Mikuláš
  - Research Site, Prešov
  - Research Site, Rimavská Sobota
  - Research Site, Ružomberok
  - Research Site, Trenčín
  - Research Site, Zvolen
- South Africa (8):
  - Research Site, Lyttleton, Centurion
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Cape Town, South Africa
  - Research Site, Durban, South Africa
  - Research Site, eMkhomazi, South Africa
  - Research Site, Durbanville
  - Research Site, eManzimtoti
  - Research Site, Pretoria
- Ukraine (8):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Vinytsa
  - Research Site, Zaporizhzhya

REFERENCES:
- [Derived] Bateman ED, O'Brien C, Rugman P, Luke S, Ivanov S, Uddin M. Efficacy and safety of the CRTh2 antagonist AZD1981 as add-on therapy to inhaled corticosteroids and long-acting beta2-agonists in patients with atopic asthma. Drug Des Devel Ther. 2018 May 4;12:1093-1106. doi: 10.2147/DDDT.S147389. eCollection 2018. PMID 29765200

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1144 participants were randomized. The first participant was enrolled on 19 October 2010 and the last participant completed the study on 16 February 2012.
Pre-assignment Details: Participants were screened for a period of 31 days out of which 17 days for enrollment and 2 weeks for run-in period.
Groups:
- AZD1981 400 mg: AZD1981 400 mg twice daily
- AZD1981 200 mg: AZD1981 200 mg once daily
- AZD1981 100 mg: AZD1981 100 mg twice daily
- AZD1981 80 mg: AZD1981 80 mg once daily
- AZD1981 40 mg: AZD1981 40 mg twice daily
- AZD1981 10 mg: AZD1981 10 mg twice daily
- Placebo: Placebo
Period: Overall Study
Arm/Group | AZD1981 400 mg | AZD1981 200 mg | AZD1981 100 mg | AZD1981 80 mg | AZD1981 40 mg | AZD1981 10 mg | Placebo
Started | 164 | 161 (Two participants did not receive study treatment) | 166 (Two participants did not receive study treatment) | 164 | 163 (One participant excluded due to Good Clinical Practice (GCP) violation at centre 4323) | 163 | 163 (Two participants excluded due to Good Clinical Practice (GCP) violation at centre 4323)
Completed | 148 | 146 | 153 | 152 | 149 | 144 | 142
Not Completed | 16 | 15 | 13 | 12 | 14 | 19 | 21
Not completed — Adverse Event | 3 | 2 | 4 | 4 | 4 | 2 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Development of study withdrawal criteria | 3 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Eligibility criteria not fulfilled | 5 | 8 | 2 | 5 | 5 | 9 | 6
Not completed — Withdrawal by Subject | 3 | 3 | 4 | 1 | 1 | 5 | 6
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Other | 1 | 1 | 3 | 0 | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Three patients (1 in the AZD1981 40 mg bid group and 2 in the placebo group) randomized at a Japanese centre were excluded from the analyses due to Good Clinical Practice violations identified after study completion.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1981 400 mg | AZD1981 200 mg | AZD1981 100 mg | AZD1981 80 mg | AZD1981 40 mg | AZD1981 10 mg | Placebo | Total
Number analyzed (Participants) | 164 | 161 | 166 | 164 | 162 | 163 | 161 | 1141
Age Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (13.98) | 46.7 (12.84) | 46.4 (14.65) | 45.4 (13.22) | 46.3 (13.15) | 44.5 (13.76) | 45.7 (13.50) | 45.9 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 82 | 87 | 78 | 82 | 80 | 76 | 561
  Male | 88 | 79 | 79 | 86 | 80 | 83 | 85 | 580
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 117 | 115 | 120 | 119 | 121 | 113 | 119 | 824
  Black or African American | 5 | 6 | 5 | 2 | 1 | 3 | 4 | 26
  Asian | 27 | 26 | 29 | 32 | 25 | 32 | 24 | 195
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 14 | 14 | 12 | 11 | 14 | 15 | 14 | 94
Time since asthma diagnosis [Mean (Standard Deviation); unit: Years] | 18.6 (13.87) | 18.5 (14.25) | 18.6 (14.74) | 18.3 (13.04) | 18.0 (14.35) | 17.3 (12.40) | 17.5 (13.27) | 18.1 (13.70)
Smoking status [Number; unit: Participants]
  Former smoker | 25 | 24 | 14 | 21 | 26 | 19 | 15 | 144
  Never | 139 | 137 | 152 | 143 | 136 | 144 | 146 | 997
Pre-bronchodilator FEV1 percentage of predicted normal (PN) at randomization [Mean (Standard Deviation); unit: Percentage of predicted normal] | 70.03 (10.544) | 68.86 (11.580) | 68.86 (11.774) | 68.56 (12.186) | 67.28 (11.732) | 69.06 (12.132) | 68.52 (11.319) | 68.73 (11.615)
Total daily dose of inhaled glucocorticosteroids (ICS) [Mean (Full Range); unit: µg] | 406.31 [125.0 to 1000.0] | 399.75 [100.0 to 1000.0] | 413.70 [125.0 to 1000.0] | 396.46 [150.0 to 500.0] | 405.56 [160.0 to 1000.0] | 418.19 [125.0 to 1000.0] | 410.99 [160.0 to 1000.0] | 407.30 [100.0 to 1000.0]

OUTCOME MEASURES:

1. Primary Outcome: Pre-bronchodilator FEV1 at the Clinic
Description: Change from baseline: treatment period average minus baseline. Treatment period average defined as the mean of all available data during randomized treatment that occurred on or prior to treatment failure. Treatment failure defined as worsening asthma symptoms resulting in increased dose of inhaled corticosteroid.
Time Frame: Twelve week treatment period
Population: The full analysis set consist of all randomized participants who received at least one dose of study medication and contributed sufficient data for at least the primary or secondary efficacy endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- Arm 1 - AZD1981 400 mg: AZD1981 400 mg twice daily
- Arm 2 - AZD1981 200 mg: AZD1981 200 mg once daily
- Arm 3 - AZD1981 100 mg: AZD1981 100 mg twice daily
- Arm 4 - AZD1981 80 mg: AZD1981 80 mg once daily
- Arm 5 - AZD1981 40 mg: AZD1981 40 mg twice daily
- Arm 6 - AZD1981 10 mg: AZD1981 10 mg twice daily
- Arm7-Placebo: Placebo
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm7-Placebo
Number analyzed (Participants) | 160 | 156 | 162 | 159 | 158 | 157 | 154
Liters | 0.16 [0.10 to 0.21] | 0.19 [0.14 to 0.25] | 0.19 [0.13 to 0.24] | 0.15 [0.10 to 0.21] | 0.20 [0.15 to 0.26] | 0.15 [0.10 to 0.21] | 0.14 [0.08 to 0.19]

2. Secondary Outcome: Morning and Evening PEF
Description: Change from baseline: treatment period average minus baseline. Treatment period average defined as the mean of all available morning (evening) PEF during randomized treatment that occurred on or prior to treatment failure. Treatment failure defined as worsening asthma symptoms resulting in increased dose of inhaled corticosteroid.
Time Frame: Twelve week treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/minute
Groups:
- Arm 7-Placebo: Placebo
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm 7-Placebo
Number analyzed (Participants) | 163 | 159 | 164 | 164 | 161 | 162 | 160
Liters/minute
  Morning PEF | 5.80 [-0.99 to 12.59] | 0.60 [-6.26 to 7.47] | 4.70 [-2.06 to 11.46] | 0.06 [-6.70 to 6.82] | 9.36 [2.54 to 16.18] | 0.36 [-6.44 to 7.16] | -1.65 [-8.49 to 5.18]
  Evening PEF | 0.78 [-6.15 to 7.72] | -1.51 [-8.54 to 5.52] | -0.20 [-7.11 to 6.71] | -5.34 [-12.25 to 1.57] | 7.20 [0.21 to 14.19] | -2.93 [-9.88 to 4.02] | 0.27 [-6.69 to 7.24]

3. Secondary Outcome: Asthma Control Questionnaire 5-item (ACQ5)
Description: The ACQ5 consists of 5 questions, each assessed on a scale from 0-6, where 0 represents good asthma control and 6 represents poor asthma control. The overall score is the mean of the responses. The minimal important difference is defined as a change in score of 0.5. Change from baseline: treatment period average minus baseline.
Time Frame: Twelve week treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on scale
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm7-Placebo
Number analyzed (Participants) | 156 | 153 | 160 | 157 | 155 | 152 | 148
Scores on scale | -0.88 [-1.00 to -0.76] | -0.88 [-1.01 to -0.76] | -0.87 [-0.99 to -0.75] | -0.90 [-1.03 to -0.78] | -0.98 [-1.10 to -0.86] | -0.83 [-0.96 to -0.71] | -0.78 [-0.91 to -0.66]

4. Secondary Outcome: Adverse Events
Description: Number of participants who had at least one adverse event during the randomized treatment period
Time Frame: Twelve week treatment period
Population: All randomized participants who received at least one dose of study medication and from whom any data after randomization was available
Measure: Number; unit: Participants
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm7-Placebo
Number analyzed (Participants) | 164 | 159 | 164 | 164 | 163 | 163 | 163
Participants | 46 | 46 | 46 | 40 | 49 | 56 | 49

5. Secondary Outcome: Number of Participants With at Least One Severe Asthma Exacerbation
Description: Severe asthma exacerbation defined as deterioration in asthma leading to either hospitalization/emergency room treatment or oral glucocorticosteroid treatment for at least 3 days
Time Frame: Twelve week treatment period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm7-Placebo
Number analyzed (Participants) | 164 | 159 | 164 | 164 | 162 | 163 | 161
Participants | 4 | 3 | 7 | 7 | 5 | 6 | 5

6. Secondary Outcome: Number of Participants With at Least One Treatment Failure
Description: Treatment failure is defined as a clinical need for additional inhaled corticosteroid use as judged by the investigator based on evaluations at the clinic.
Time Frame: Twelve week treatment period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm7-Placebo
Number analyzed (Participants) | 164 | 159 | 164 | 164 | 162 | 163 | 161
Participants | 4 | 9 | 3 | 8 | 10 | 12 | 12

7. Secondary Outcome: Number of Participants With Well-controlled Asthma (ACQ5<=0.75)
Description: The ACQ5 consists of 5 questions, each assessed on a scale from 0-6, where 0 represents good asthma control and 6 represents poor asthma control. The overall score is the mean of the responses. Well-controlled asthma is defined as ACQ5<=0.75 at the end of the 12-week treatment period.
Time Frame: Twelve week treatment period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm7-Placebo
Number analyzed (Participants) | 164 | 159 | 164 | 164 | 162 | 163 | 161
Participants | 34 | 33 | 34 | 34 | 36 | 30 | 19

8. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ(S))
Description: The AQLQ(S) consists of 32 questions, each assessed on a scale from 1-7, with higher values indicating better health-related quality of life. Overall scores are calculated from the means of the individual scores. The minimal important difference is a change in score of 0.5. Change from baseline: treatment period average minus baseline.
Time Frame: Twelve week treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm7-Placebo
Number analyzed (Participants) | 156 | 152 | 160 | 157 | 155 | 152 | 148
Score on scale | 0.73 [0.60 to 0.85] | 0.73 [0.61 to 0.86] | 0.75 [0.63 to 0.87] | 0.80 [0.68 to 0.92] | 0.82 [0.69 to 0.94] | 0.72 [0.59 to 0.84] | 0.65 [0.53 to 0.78]

9. Secondary Outcome: Asthma Symptom Score
Description: Asthma symptoms, measured in the morning and evening, based on a scale from 0-3 with higher scores indicating more severe asthma symptoms. Total asthma symptom score (0-6) is calculated by taking the sum of the morning and evening scores. Change from baseline: treatment period average minus baseline.
Time Frame: Twelve week treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm7-Placebo
Number analyzed (Participants) | 164 | 158 | 164 | 164 | 162 | 163 | 160
Score on scale | -0.30 [-0.42 to -0.18] | -0.26 [-0.38 to -0.14] | -0.28 [-0.40 to -0.16] | -0.33 [-0.45 to -0.21] | -0.34 [-0.46 to -0.22] | -0.30 [-0.42 to -0.17] | -0.27 [-0.39 to -0.15]

10. Secondary Outcome: Total Reliever Medication Use
Description: Reliever medication use (number of inhalations), measured in the morning and evening. Total reliever medication use is calculated by taking the sum of the number of daytime and evening inhalations of reliever medication. Change from baseline: treatment period average minus baseline.
Time Frame: Twelve week treatment period
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of inhalations
Arm/Group | Arm 1 - AZD1981 400 mg | Arm 2 - AZD1981 200 mg | Arm 3 - AZD1981 100 mg | Arm 4 - AZD1981 80 mg | Arm 5 - AZD1981 40 mg | Arm 6 - AZD1981 10 mg | Arm7-Placebo
Number analyzed (Participants) | 164 | 158 | 164 | 164 | 162 | 163 | 160
Number of inhalations | -0.51 [-0.72 to -0.31] | -0.22 [-0.43 to -0.01] | -0.38 [-0.58 to -0.17] | -0.39 [-0.59 to -0.18] | -0.37 [-0.58 to -0.17] | -0.37 [-0.58 to -0.17] | -0.35 [-0.56 to -0.15]

ADVERSE EVENTS:
Arm/Group | AZD1981 400 mg | AZD1981 200 mg | AZD1981 100 mg | AZD1981 80 mg | AZD1981 40 mg | AZD1981 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/164 | 1/159 | 3/164 | 1/164 | 0/163 | 0/163 | 1/163
Other Adverse Events (participants affected / at risk) | 12/164 | 23/159 | 22/164 | 21/164 | 20/163 | 32/163 | 21/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1981 400 mg (N=164) | AZD1981 200 mg (N=159) | AZD1981 100 mg (N=164) | AZD1981 80 mg (N=164) | AZD1981 40 mg (N=163) | AZD1981 10 mg (N=163) | Placebo (N=163)
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1981 400 mg (N=164) | AZD1981 200 mg (N=159) | AZD1981 100 mg (N=164) | AZD1981 80 mg (N=164) | AZD1981 40 mg (N=163) | AZD1981 10 mg (N=163) | Placebo (N=163)
Nasopharyngitis (Infections and infestations) | 4 | 10 | 7 | 9 | 5 | 10 | 6
Bronchitis (Infections and infestations) | 1 | 4 | 2 | 1 | 5 | 5 | 5
Pharyngitis (Infections and infestations) | 2 | 2 | 4 | 4 | 3 | 3 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 3 | 5 | 4
Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 5 | 2
Headache (Nervous system disorders) | 2 | 7 | 7 | 4 | 3 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 3 | 2 | 4 | 3
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less